CLINICAL TRIAL: NCT06963801
Title: Developing Pregnancy-specific Dialectical Behavior Therapy Skills to Promote Multigenerational Mental Health
Brief Title: DBT-P Treatment Study
Acronym: REACH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Oregon (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00116252; R61MH138444 (NIH)
Record Dates: First submitted 2025-04-30; First posted 2025-05-09 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-04

CONDITIONS: Emotion Dysregulation
Keywords: Emotion dysregulation; Pregnancy; Maternal health; RSA; Coping; Stress; DBT-P; Moms2B

STUDY DESIGN:
Intervention Model Description: Two groups: control group is assessment only and treatment group is DBT-P group sessions (emotional skills regulation groups). Groups stratified based on gestational age (14-20 weeks vs 21-27 weeks) as well as race and ethnicity.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The Clinical Research Coordinators collecting the data and conducting semi-structured emotion regulation interview.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moms2B (Active Comparator): Moms2B is an established group-based intervention for pregnant women focused on enhancing social support and improving nutrition. Participants will receive 3 sessions using this established assessment only treatment plan as well as complete surveys and clinical interviews assessing stress, coping strategies and emotions. Resting heart rate data as well as heart rate data post stimulus to be assessed.
  Interventions: Behavioral: Moms2B
- DBT-P (Experimental): DBT-P is a Dialectical Behavior Therapy skills group adapted for pregnant people. Participants will receive weekly DBT-P group sessions for 10 weeks where they learn skills to: (1) enhance self-awareness; (2) improve ability to manage crises; (3) decrease negative emotions and increase positive emotions; (4) improve your relationships and self-respect; they will also complete homework as part of the group participation as well as complete daily diary cards that will ask about their mood and any thoughts of self-harm .
  Completion of surveys and clinical interviews assessing stress, coping strategies and emotions are included; resting heart rate data as well as heart rate data post stimulus to be assessed.
  Interventions: Behavioral: Moms2B; Behavioral: DBT-P

INTERVENTIONS:
Behavioral: Moms2B — An established group-based pregnancy program focusing on improving nutrition, social, and medical support.
Behavioral: DBT-P — An emotional skills group where emotion regulation skills are taught in the context of the pregnancy and expected life with an infant.
  Arms: DBT-P

SUMMARY:
The goal of this study is to find out if improving emotion regulation skills use during pregnancy reduces maternal stress and improves heart rate.

The main questions it aims to answer are:

* Does improving emotion regulation skills during pregnancy reduce stress and improve the ability to cope?
* How is a participant's heart rate affected by their ability to control their emotions during pregnancy?

Researchers will test the hypothesis that dialectical behavior therapy skills groups (DBT-P) will improve emotion regulation skills use as well as heart rate.

Participants will:

* Visit the clinic for 3 sessions at the beginning, middle and end of their pregnancy.
* Compete surveys and interviews asking about their thoughts, feelings and how they cope with emotions.
* Have their heart rate taken.
* If assigned to the investigational group, they will complete weekly remote emotion regulation skills groups for 10 weeks and complete daily diary cards that ask about mood and any thoughts of self-harm.
* Optional Element: Complete a 20-30min infant neurobehavior exam (NNNS exam) after delivery.

DETAILED DESCRIPTION:
The investigators' observational research with mothers with emotion dysregulation and their infants shows that poor emotion regulation skill use is a mechanism that likely confers risk for self-injurious thoughts and behaviors, depression, and anxiety in the mother and neurobehavioral and co-regulatory challenges in the infant. Emotion dysregulation is an impairing, early-emerging, transdiagnostic vulnerability factor that has intergenerational implications. Treatments have been developed for non-pregnant adults with emotion dysregulation but these are costly, time-intensive, and do not address the unique needs of pregnant people, highlighting an unmet therapeutic need. Through this innovative intervention, researchers will test whether targeting emotion regulation skills use during pregnancy will both improve postpartum emotion regulation, newborn neurobehavior, and mother-infant co-regulation. Early identification of the mechanisms implicated in risk. The researchers will deliver 10 weeks of DBT skills classes selected and adapted to meet the unique needs of pregnancy (DBT-P). The goal of this work is to improve perinatal mental health trajectories.

The premise of this study-that improving emotion regulation in pregnancy may disrupt intergenerational transmission of psychopathology-is informed by our research over the past two decades, including several NIH awards (R01MH119070, R01MH132210, R01DA049755, R21MH1090777, F31MH074196). The investigator' data reveal that maternal emotion dysregulation confers risk for mother. The research also shows that resting respiratory sinus arrhythmia (RSA), a physiological index of emotion dysregulation, can be improved via intervention in non-pregnant adults. The investigators propose that DBT-P will increase emotion regulation skills use or increase RSA in the mother (target engagement) leading to significant reductions in her emotion dysregulation prior to birth.

The primary study objectives are to recruit 100 pregnant women with high emotion dysregulation to receive either: (1) dialectical behavior therapy skills groups or an Assessment only control; and (2) to evaluate whether the treatment improved emotion regulation skills use as well as respiratory sinus arrhythmia.

ELIGIBILITY:
Inclusion Criteria:

* Emotion dysregulation score of 88 or above
* At least 12 weeks pregnant
* Singleton Pregnancy
* Fluent in English

Exclusion Criteria:

* Active psychosis
* Drug or alcohol use disorder during pregnancy
* High risk of an imminent suicide attempt
* Significant health complications (e.g., cancer)
* Illiterate and/or unable to independently complete and comprehend written measures

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2026-10-05 (Estimated); Study Completion 2026-10-19 (Estimated)

PRIMARY OUTCOMES:
Difficulties in Emotion Regulation Scale (DERS) | Baseline (Week 0), mid-treatment (Week 5), and post-treatment (Week 10)
  The DERS is a 36-item measure scored on a 5-point Likert Scale. DERS scores range from 36-180 and enrollment in this study requires a baseline total DERS score of ≥88 which indicate greater difficulties in emotion regulation.
Respiratory Sinus Arrhythmia (RSA) | Baseline (Week 0), mid-treatment (Week 5), and post-treatment (Week 10)
  RSA is a peripheral index of parasympathetic nervous system influences on cardiac activity and is measured as the variability in heart rate that coincides with respiration.

SECONDARY OUTCOMES:
Percent of participation | Baseline (Week 0), mid-treatment (Week 5), and post-treatment (Week 10)
  Feasibility of the assessment schedule will include the percent of participation at all timepoints.
Percent of missing data | Baseline (Week 0), mid-treatment (Week 5), and post-treatment (Week 10)
  Feasibility of the assessment schedule will include the percent of missing data at all time points.
Recruitment rates | Baseline (Week 0), mid-treatment (Week 5), and post-treatment (Week 10)
  Feasibility of the intervention will be assessed by evaluating recruitment rates.
Reasons for refusal | Baseline (Week 0), mid-treatment (Week 5), and post-treatment (Week 10)
  Feasibility of the intervention will be assessed by evaluating reasons for refusal. Collection of reasons for refusal to be obtained via subject self-report at each individual timepoint; expected attendance for 85% of sessions.
Intervention adherence | Baseline (Week 0), mid-treatment (Week 5), and post-treatment (Week 10)
  Feasibility of the intervention will be assessed by evaluating intervention adherence. Weekly assessment of intervention adherence conducted by clinicians based on subject completion of required homework assignments, daily diary entries and group session attendance.
Number of women who complete all sessions | Baseline (Week 0), mid-treatment (Week 5), and post-treatment (Week 10)
  Feasibility will be assessed by how many women completed all sessions.
Number of interventionists who can self-monitor for fidelity, assessed by watching segments of video-recorded sessions | Baseline (Week 0), mid-treatment (Week 5), and post-treatment (Week 10)
  Feasibility will be assessed by whether the interventionist can self-monitor for fidelity.
Participation rates | Post-treatment (Week 10)
  Acceptability will be assessed by participation rates.
Participant satisfaction with the intervention assessed by the Client Satisfaction Questionnaire | Post-treatment (Week 10)
  Acceptability will be assessed by measuring participant satisfaction with the intervention (including completion of the intervention) using the Client Satisfaction Questionnaire. Scores are summed across items once. Items 2, 4, 5, and 8 are reverse scored. Total scores range from 8 to 32, with the higher number indicating greater satisfaction.
Telehealth acceptability specific to DBT skills training | Post-treatment (Week 10)
  A 41-item original survey developed by DBT experts in the United States and Australia to measure participants' satisfaction with DBT delivered through telehealth. Items designed to assess relevance of care experience on a 5-pt scale from Not Relevant to Very Relevant. Responses anonymized and qualitative free-text fields provided for recommendations and comments for changes or improvements.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Conradt, PhD, Principal Investigator — Duke University; Andrada Neacsiu, PhD, Principal Investigator — Duke University; Sheila Crowell, PhD, Principal Investigator — University of Oregon
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No